CLINICAL TRIAL: NCT03973983
Title: Comparison of Ultrasound-guided Transgluteal and Finger-guided Transvaginal Pudendal Nerve Block Techniques: Which One is More Effective?
Brief Title: Comparison of Ultrasound-guided Transgluteal and Finger-guided Transvaginal Pudendal Nerve Block Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hande Gurbuz, Principal Investigator, Derince Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1234-5765
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Neuralgia; Pudendal Nerve; Pudendal Nerve Block
Keywords: neuralgia; pudendal nerve; pudendal nerve block; therapeutic local anaesthesia; transvaginal
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided pudendal nerve injection group (Experimental): Patients who received Ultrasound-guided pudendal nerve injections
  Interventions: Procedure: Ultrasound-guided transgluteal pudendal nerve injection (TG-PNI)
- Finger-guided pudendal nerve injection group (Experimental): Patients who received Finger-guided pudendal nerve injections
  Interventions: Procedure: Finger-guided transvaginal pudendal nerve injection (TV-PNI)

INTERVENTIONS:
Procedure: Ultrasound-guided transgluteal pudendal nerve injection (TG-PNI) — Ultrasound-guided transgluteal pudendal nerve local anesthetic injections
  Arms: Ultrasound-guided pudendal nerve injection group
Procedure: Finger-guided transvaginal pudendal nerve injection (TV-PNI) — Finger-guided transvaginal pudendal nerve local anesthetic injections
  Arms: Finger-guided pudendal nerve injection group

SUMMARY:
Pudendal neuralgia (PN) is a painful and disabling condition, which reduces the quality of life as well. Pudendal nerve injections are essential for the diagnosis and the management of PN. The purpose of this study was to compare the effectiveness of finger-guided transvaginal pudendal nerve injection (TV-PNI) technique and the US-guided transgluteal pudendal nerve injection (TG-PNI) technique.

DETAILED DESCRIPTION:
Pudendal neuralgia (PN) is a painful neuropathic condition for which current prevalence is unknown due to often going under-recognized by gynecologists. Pudendal neuralgia typically presents as unilateral severe sharp and burning pain, numbness, or paranesthesia on the anatomic pathways of the pudendal nerve. The most common causes for PN include pudendal nerve injury during vaginal procedures, stretching and compression of the pudendal nerve during vaginal delivery, and prolonged sitting position.

As in many neuropathic syndromes, there is currently no gold standard diagnostic test for assessing PN. In 2006, the Nantes criteria were described by a multidisciplinary working party to describe the clinical diagnostic criteria, and a standard approach was created for PN diagnosis. According to the Nantes criteria, patients should fulfil all five essential criteria without meeting any of the exclusion criteria. The five essential diagnostic criteria were defined as, 1: pain in the anatomic territory of the pudendal nerve, 2: that is worsened by sitting, 3: the patient is not woken at night by the pain, 4: no objective sensory loss on clinical examination, and 5: positive anesthetic pudendal nerve block.

Pudendal nerve infiltration (PNI), which was defined as an essential step, is performed for diagnostic purposes and as an important treatment modality in patients with PN. This approach aims for long-term relief of pain, as in all forms of nerve entrapment syndromes, by treating a possible inflammatory component, it also provides neuroprotection to the central nervous system and reduces spontaneous ectopic activity of the affected nerve.

Image-guided or finger-guided PNIs can be performed according to the experience of the physician, adequate equipment presence, and patient choice. The pudendal nerve is situated in the deepest area in the pelvis and it makes the PNI technically difficult if transperineal or transgluteal approaches are preferred. For this reason, it usually requires imaging guidance to target the injection site such as ultrasound, computed tomography, fluoroscopy, and magnetic resonance.

Ultrasound-guided transgluteal (TG) PNI has been described to reach the pudendal nerve in the plane between the sacrotuberous and sacrospinous ligaments. This technique has many advantages such as visualization of the substantial structures (pudendal artery and the sciatic nerve) without radiation exposure it enables real-time images. However, finger-guided transvaginal (TV) PNI should be kept in mind as a PNI option with the advantages of familiarity for gynecologists and obstetricians as an essential part of obstetric anesthesia. Finger-guided blocks in women are easily performed via a vaginal approach by palpation the ischial spines and the injection is targeted slightly medially and posteriorly to the ischial spines.

Over the past 20 years, studies have described the PNI techniques, but a limited number of studies have compared the efficacy of image-guided PNI techniques. To the best of our knowledge, there are no studies comparing the finger-guided TV-PNI and US-guided TG-PNI for the evaluation of pain relief in patients with PN. We hypothesized that the finger-guided TV technique is effective as US-guided TG-PNI when performed to relieve pain in patients with PN. The primary outcome of the present study was to evaluate the changes of mean VAS scores based on the mean daily maximum pain intensity score during the week before day 0 (D0), day 7 (D7), day 21 (D21), and day 180 (D180). Secondly, the post-block complication rate was evaluated in overall blocks. Secondary outcome included the comparison of the success rates of both two techniques (from D0 to D180).

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnostic pudendal nerve injection (PNI)

Exclusion Criteria:

* Negative diagnostic pudendal nerve injection (PNI)
* Virgin
* Sexual inactive

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 180 days
  Post-injection pain scores (while sitting, while/after intercourse and pain in the region from the anus to the clitoris) (ward) Pain scores were assessed with a 10-cm Visual Analogue Scale (VAS) (with 0 = no pain and 10 = the worst imaginable pain)

SECONDARY OUTCOMES:
Block success | 180 days
  The comparison of the success rates of both two techniques (finger guided TV-PNI vs ultrasound guided TG-PNI) Improvement of more than 50% of the initial pain VAS scores at 6 months after the PNIs completed was considered as clinical success.

CONTACTS AND LOCATIONS:
Locations (1):
- Hande G. Aytuluk, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roth TM. Management of persistent groin pain after transobturator slings. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Nov;18(11):1371-3. doi: 10.1007/s00192-007-0365-1. Epub 2007 Apr 13. PMID 17431534
- [Background] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Background] Vancaillie T, Eggermont J, Armstrong G, Jarvis S, Liu J, Beg N. Response to pudendal nerve block in women with pudendal neuralgia. Pain Med. 2012 Apr;13(4):596-603. doi: 10.1111/j.1526-4637.2012.01343.x. Epub 2012 Mar 5. PMID 22390343
- [Result] Ramsden CE, McDaniel MC, Harmon RL, Renney KM, Faure A. Pudendal nerve entrapment as source of intractable perineal pain. Am J Phys Med Rehabil. 2003 Jun;82(6):479-84. PMID 12820792
- [Result] Labat JJ, Riant T, Robert R, Amarenco G, Lefaucheur JP, Rigaud J. Diagnostic criteria for pudendal neuralgia by pudendal nerve entrapment (Nantes criteria). Neurourol Urodyn. 2008;27(4):306-10. doi: 10.1002/nau.20505. PMID 17828787
- [Result] Kastler A, Puget J, Tiberghien F, Pellat JM, Krainik A, Kastler B. Dual Site Pudendal Nerve Infiltration: More than Just a Diagnostic Test? Pain Physician. 2018 Jan;21(1):83-90. PMID 29357337
- [Result] Fanucci E, Manenti G, Ursone A, Fusco N, Mylonakou I, D'Urso S, Simonetti G. Role of interventional radiology in pudendal neuralgia: a description of techniques and review of the literature. Radiol Med. 2009 Apr;114(3):425-36. doi: 10.1007/s11547-009-0371-0. Epub 2009 Mar 10. English, Italian. PMID 19277838